CLINICAL TRIAL: NCT02710929
Title: A Genome-wide Association Study on the Endophenotype of Spatial Working Memory in Attention Deficit Hyperactivity Disorder
Brief Title: A Genome-wide Association Study on the Endophenotype of Spatial Working Memory in ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412157RINA
Record Dates: First submitted 2016-03-13; First posted 2016-03-17 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Attention-deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 15 ml blood will be withdrawn from the subjects (one heparin-rinsed tube for cell culture, one EDTA rinsed tube for DNA extraction)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD group: Subjects with clinical diagnosis of ADHD according to the DSM-IV criteria
- TD group: Typically development controls without lifetime diagnosis with ADHD

SUMMARY:
Specific Aims:

1. To find the genetic variations associated with spatial working memory performance in patients with ADHD by using genome-wide association studies (GWAS);
2. To find the genetic variations associated with spatial working memory performance in healthy subjects by using GWAS;
3. To recruit a validation sample and to replicate the findings from the initial GWAS;
4. To test whether genetic variations significantly associated with spatial working memory are also associated with ADHD.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD), characterized by inattention, hyperactivity and impulsivity, is an early onset, highly heritable, clinically heterogeneous, long-term impairing disorder with tremendous impact on individuals, families, and societies. Our research team has conducted a series of biological studies on spatial working memory deficits of ADHD, and substantial evidence has suggested spatial working memory deficits as the important neuropsychological biomarker with translational values and favorable endophenotypic properties for ADHD. Despite the abundance of molecular genetic studies on ADHD, the genetic etiologies of ADHD have been non-conclusive. Because genetic studies on endophenotypes can offer more information on genetic and brain process, endophenotypic approach can efficiently enhance the statistical power and make genome-wide association studies (GWAS) applicable in much smaller sample. To date, there has been no GWAS study on spatial working memory deficits of ADHD.

This is a 3-year project. Our previous studies have collected blood samples and spatial working memory data of 382 patients with ADHD and 150 healthy subjects. In this 3-year project, we will recruit 232 healthy subjects, aged 7-18 years. The measures include (1) interviews for psychopathology (K-SADS-E), (2) questionnaires to measures ADHD symptoms (SNAP-IV), and (3) neuropsychological tests: Spatial Working Memory task of the CANTAB. In the first year, a case-only GWAS on spatial working memory (n = 254) will be conducted. In the second year, a control-only GWAS on spatial working memory (n = 254) will be conducted. In the third year, findings from the initial two GWAS will be replicated in a validation sample composed of 128 patients with ADHD and 128 healthy controls.

By careful calculation, a sample size of 382 ADHD subjects will provide adequate power to detect genome-wide significant genetic variations and replicate the findings in an independent validation sample. We anticipate to identify the relationship between genetic variations of ADHD and the endophenotype of spatial working memory. Our findings will significantly contribute to our understanding of the pathophysiological mechanisms of ADHD, especially the pathological pathway from genes, through endophenotype, to behavioral phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without any current or lifetime DSM-IV psychiatric disorders based on the K-SADS-E interviews.

Exclusion Criteria:

* Participants who had any past or current medical or neurological illness, who currently took psychotropic medication, or whose intelligence quotient (IQ) score was less than 80 were excluded.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The existing sample is composed of 382 children withADHD and 150 healthy subjects. We plan to recruit additional 232 healthy subjects (104 in the first year; 128 in the second year), aged 7 to 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Psychiatric interview | 1 hour
  Subjects will be interviewed by Chinese Version of the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E)

SECONDARY OUTCOMES:
Spatial working memory | 30 minutes
  Subjects will be assessed by the Cambridge Neuropsychological Test Automated Battery (CANTAB)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yung Shang, MD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No